CLINICAL TRIAL: NCT02459899
Title: A Phase 2b, Dose-ranging, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study in Patients With Type 1 Diabetes Mellitus Who Have Inadequate Glycemic Control With Insulin Therapy
Brief Title: Dose-ranging Study in Patients With Type 1 Diabetes Mellitus
Acronym: inTandem4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX4211.1-206-T1DM; LX4211.206 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Two placebo-matching sotagliflozin tablets, once daily, orally for 12 weeks.
  Interventions: Drug: Placebo
- Sotagliflozin 75 mg (Experimental): Sotagliflozin 75 mg (one 75 mg tablet and one placebo tablet), once daily, orally for 12 weeks.
  Interventions: Drug: Placebo; Drug: Sotagliflozin
- Sotagliflozin 200 mg (Experimental): Sotagliflozin 200 mg (one 200 mg tablet and one placebo tablet), once daily, orally for 12 weeks.
  Interventions: Drug: Placebo; Drug: Sotagliflozin
- Sotagliflozin 400 mg (Experimental): Sotagliflozin 400 mg (two 200 mg tablets), once daily, orally for 12 weeks.
  Interventions: Drug: Sotagliflozin

INTERVENTIONS:
Drug: Placebo — Placebo, once daily, before the first meal of the day
  Arms: Placebo; Sotagliflozin 200 mg; Sotagliflozin 75 mg
Drug: Sotagliflozin — Sotagliflozin,once daily, before the first meal of the day
  Arms: Sotagliflozin 200 mg; Sotagliflozin 400 mg; Sotagliflozin 75 mg

SUMMARY:
The primary objective of this study was to define the dose leading to desirable efficacy, as measured by the change in hemoglobin A1C (A1C) between Baseline and Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Participant had given written informed consent to participate in the study in accordance with local regulations.
* Adult participants 18 years and older with a diagnosis of type 1 diabetes mellitus (T1D) made at least 1 year prior to informed consent.
* Participants were being treated with insulin or insulin analog delivered via continuous subcutaneous insulin infusion (CSII) or multiple daily injection (MDI).
* At the Screening Visit, A1C had to be between 7.0% and 10.0%.
* Females of childbearing potential had to use an adequate method of contraception and have a negative pregnancy test.

Exclusion Criteria:

* Use of antidiabetic agent other than insulin or insulin analog at the time of screening.
* Use of sodium-glucose cotransporter (SGLT) inhibitors within 8 weeks prior to screening.
* Chronic systemic corticosteroid use.
* Type 2 diabetes mellitus (T2DM), or severely uncontrolled T1D as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (17):
- United States (17):
  - Lexicon Investigational Site, Concord, California
  - Lexicon Investigational Site, Ventura, California
  - Lexicon Investigational Site, Denver, Colorado
  - Lexicon Investigational Site, Jacksonville, Florida
  - Lexicon Investigational Site, Miami, Florida
  - Lexicon Investigational Site, Springfield, Illinois
  - Lexicon Investigational Site, Metairie, Louisiana
  - Lexicon Investigational Site, Auburn, Maine
  - Lexicon Investigational Site, Rockville, Maryland
  - Lexicon Investigational Site, Great Falls, Montana
  - Lexicon Investigational Site, Omaha, Nebraska
  - Lexicon Investigational Site, High Point, North Carolina
  - Lexicon Investigational Site, Columbus, Ohio
  - Lexicon Investigational Site, San Antonio, Texas
  - Lexicon Investigational Site, Salt Lake City, Utah
  - Lexicon Investigational Site, Chesapeake, Virginia
  - Lexicon Investigational Site, Manassas, Virginia

REFERENCES:
- [Derived] Baker C, Wason S, Banks P, Sawhney S, Chang A, Danne T, Gesty-Palmer D, Kushner JA, McGuire DK, Mikell F, O'Neill M, Peters AL, Strumph P. Dose-dependent glycometabolic effects of sotagliflozin on type 1 diabetes over 12 weeks: The inTandem4 trial. Diabetes Obes Metab. 2019 Nov;21(11):2440-2449. doi: 10.1111/dom.13825. Epub 2019 Aug 1. PMID 31264767

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 17 centers in the United States from 10 July 2015 to 26 August 2016.
Pre-assignment Details: 207 participants were screened and 141 participants with Type 1 diabetes mellitus who had inadequate glycemic control with insulin therapy alone, were randomized equally into four treatment groups: sotagliflozin 75 milligrams (mg), sotagliflozin 200 mg, sotagliflozin 400 mg or placebo.
Groups:
- Sotagliflozin 75 mg: Sotagliflozin 75 mg (one 75 mg tablet and one placebo tablet), once daily, orally, for 12 weeks.
- Sotagliflozin 200 mg: Sotagliflozin 200 mg (one 200 mg tablet and one placebo tablet), once daily, orally, for 12 weeks.
- Sotagliflozin 400 mg: Sotagliflozin 400 mg (two 200 mg tablets), once daily, orally, for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Sotagliflozin 75 mg | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Started | 36 | 35 | 35 | 35
Completed | 33 | 29 | 35 | 33
Not Completed | 3 | 6 | 0 | 2
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 1
Not completed — Non-compliance with the treatment | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-treat (mITT) population consisted of all randomly assigned participants who had taken at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sotagliflozin 75 mg | Sotagliflozin 200 mg | Sotagliflozin 400 mg | Total
Number analyzed (Participants) | 36 | 35 | 35 | 35 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (11.29) | 42.4 (12.01) | 47.0 (14.01) | 44.8 (15.36) | 45.6 (13.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 15 | 15 | 73
  Male | 15 | 13 | 20 | 20 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 4 | 3 | 0 | 7
  White | 34 | 31 | 31 | 35 | 131
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Body Weight [Mean (Standard Deviation); unit: kilograms] | 91.92 (19.681) | 79.97 (14.358) | 82.90 (17.140) | 86.95 (20.857) | 85.48 (18.557)
Daily Total Insulin Dose [Mean (Standard Deviation); unit: International units per kilogram (IU/kg)] | 0.68 (0.306) | 0.65 (0.229) | 0.70 (0.298) | 0.77 (0.409) | 0.70 (0.315)
Hemoglobin A1C (A1c) [Mean (Standard Deviation); unit: percentage of A1C] | 7.95 (0.849) | 8.00 (0.839) | 8.07 (0.926) | 8.05 (0.735) | 8.02 (0.832)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per meter square] | 31.81 (5.763) | 27.41 (5.016) | 28.01 (4.707) | 29.37 (5.849) | 29.17 (5.569)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 26.9 (13.51) | 22.2 (13.04) | 23.4 (13.17) | 24.0 (14.96) | 24.1 (13.66)
Insulin delivery method in Participants [Count of Participants; unit: Participants]
  continuous subcutaneous insulin infusion (CSII) | 19 | 18 | 18 | 18 | 73
  multiple daily injection (MDI) | 17 | 17 | 17 | 17 | 68

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C (A1C) at Week 12
Description: Baseline was defined as the last value collected prior to the first dose of double-blind study medication. Post-baseline Least Square (LS) mean values were obtained from mixed-effects model repeated measures (MMRM) model with treatment, randomization strata of insulin delivery method (continuous subcutaneous insulin infusion [CSII] or multiple daily injection [MDI]), time (study week), and a treatment-by-time interaction as fixed categorical effects, and baseline A1C-by-time interaction as a covariate.
Time Frame: Baseline to Week 12
Population: Analysis included participants from the mITT population. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percentage of A1C
Arm/Group | Placebo | Sotagliflozin 75 mg | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 33 | 29 | 35 | 33
percentage of A1C | -0.35 (0.096) | -0.60 (0.100) | -0.84 (0.095) | -0.73 (0.096)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 75 mg; Analysis was performed using MMRM model with treatment, randomization strata of insulin delivery method (CSII, MDI), time (study week), and a treatment-by-time interaction as fixed categorical effects, and Baseline A1C-by-time interaction as a covariate; Test type: Superiority; p = 0.07, MMRM — Threshold for significance < 0.05; Least squares mean difference = -0.25, 95% CI 2-sided [-0.53 to 0.02], Standard Error of Mean 0.139
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 200 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, MMRM — Threshold for significance < 0.05; Least squares mean difference = -0.48, 95% CI 2-sided [-0.75 to -0.22], Standard Error of Mean 0.135
Statistical Analysis 3: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.006, MMRM — Threshold for significance < 0.05; Least squares mean difference = -0.38, 95% CI 2-sided [-0.65 to -0.11], Standard Error of Mean 0.136

2. Secondary Outcome: Change From Baseline to Week 12 in 2-Hour Postprandial Glucose (PPG) Following the Standardized Mixed Meal
Description: A 2-hour PPG sample (plasma) was obtained 2-hours after a standardized Mixed Meal at Baseline (Day 1) and at the visit at Week 12. Post-Baseline LS mean was obtained from analysis of covariance (ANCOVA) model with treatment, randomization strata of insulin delivery method (CSII, MDI) as fixed categorical effects, and baseline postprandial glucose as a covariate.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Placebo | Sotagliflozin 75 mg | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 32 | 27 | 25 | 32
milligrams per deciliter (mg/dL) | -0.2 (12.51) | -20.5 (13.66) | -27.6 (14.16) | -49.7 (12.51)

3. Secondary Outcome: Absolute Change From Baseline in Body Weight to Week 12
Description: Baseline was defined as the last value collected prior to the first dose of double-blind study medication. Post-Baseline LS mean was obtained from MMRM model with treatment, randomization strata of insulin delivery method (CSII, MDI), time (study week), and a treatment-by-time interaction as fixed categorical effects, and baseline weight-by-time interaction as a covariate.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Placebo | Sotagliflozin 75 mg | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 33 | 29 | 35 | 33
kilograms | 1.13 (0.425) | -0.16 (0.441) | -1.24 (0.417) | -1.48 (0.422)

4. Secondary Outcome: Percent Change From Baseline in Body Weight to Week 12
Description: as for outcome 3
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Sotagliflozin 75 mg | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 33 | 29 | 35 | 33
percent change | 1.26 (0.535) | 0.11 (0.556) | -1.47 (0.531) | -1.61 (0.538)

5. Secondary Outcome: Change From Baseline to Week 12 in 24-Hour Urinary Glucose Excretion
Description: Urine was collected over 24 hours to measure Urinary Glucose Excretion at baseline, and at the end of the 12-week treatment. Post-Baseline LS mean was obtained from ANCOVA model with treatment, randomization strata of insulin delivery method (CSII, MDI) as fixed categorical effects, and Baseline urinary glucose excretion as a covariate.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: grams per day
Arm/Group | Placebo | Sotagliflozin 75 mg | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 23 | 24 | 23 | 24
grams per day | 0.2555 (10.53532) | 42.0185 (10.52465) | 57.9850 (10.51367) | 70.7058 (10.28691)

6. Secondary Outcome: Change From Baseline to Week 12 in Fasting Plasma Glucose
Description: Baseline was defined as the last value collected prior to the first dose of double-blind study medication. Post-Baseline LS mean was obtained from MMRM model with treatment, randomization strata of insulin delivery method (CSII, MDI), time (study week), and a treatment-by-time interaction as fixed categorical effects, and baseline fasting plasma glucose-by-time interaction as a covariate.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Sotagliflozin 75 mg | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 33 | 29 | 34 | 33
mg/dL | -10.8 (8.99) | -19.4 (9.55) | -19.8 (8.85) | -32.2 (8.99)

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from first dose up to 30 days after date of last dose of double-blind study treatment (up to 114 days)
Description: Analysis was performed on safety population which included all randomized participants who had received at least 1 dose of study drug.
Groups:
- Placebo: Two placebo-matching sotagliflozin tablets, once daily, orally, for 12 weeks.
Arm/Group | Placebo | Sotagliflozin 75 mg | Sotagliflozin 200 mg | Sotagliflozin 400 mg
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/35 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 1/36 | 1/35 | 1/35 | 1/35
Other Adverse Events (participants affected / at risk) | 10/36 | 5/35 | 6/35 | 4/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | Sotagliflozin 75 mg (N=35) | Sotagliflozin 200 mg (N=35) | Sotagliflozin 400 mg (N=35)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | Sotagliflozin 75 mg (N=35) | Sotagliflozin 200 mg (N=35) | Sotagliflozin 400 mg (N=35)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 4 (6) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.